CLINICAL TRIAL: NCT04259814
Title: Effect of mCIMT Casting on Speech-language Outcomes in Children With Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Sudarshan Dayanidhi, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00211104
Record Dates: First submitted 2020-02-04; First posted 2020-02-07 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Speech and Language Disorder; Cerebral Palsy; Hemiplegia; Hemiparesis
Keywords: speech delay; one-sided weakness
MeSH Terms: conditions — Speech; Language Disorders; Cerebral Palsy; Hemiplegia; Paresis; Language Development Disorders | interventions — Speech Therapy

STUDY DESIGN:
Intervention Model Description: Non-concurrent, multiple-baseline across participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Speech-Language Treatment plus mCIMT (Experimental): 4 participants
  Baseline phase: Speech-language treatment (SLT), 1 hour a day, 3 days a week. The length of the baseline phase will be staggered across subjects.
  Treatment phase: SLT combined with modified constraint-induced movement therapy(mCIMT) 1 hour a day, 3 days a week.
  Total of baseline and treatment sessions will be 20 to 30 sessions.
  Interventions: Behavioral: Speech-language therapy (SLT); Behavioral: Modified constraint-induced movement therapy (mCIMT)

INTERVENTIONS:
Behavioral: Speech-language therapy (SLT) — Age-appropriate play activities with speech-language pathologist (SLP) to elicit speech, using stimulation strategies including but not limited to recasts, expansion, parallel talk, interactive modeling, communication temptations, and phrase completions. Activities will include an age-appropriate story, pretend play (i.e., house with people, playing with a baby doll), an assembly task (i.e., building blocks, making pretend pizza), and a highly motivating, clinician-controlled activity (i.e., blowing bubbles, swing, pushing cars down a ramp).
Behavioral: Modified constraint-induced movement therapy (mCIMT) — Participants will wear a removable cast and an occupational therapist will be present during therapy to focus on facilitating play with the affected arm.

SUMMARY:
Modified constraint-induced movement therapy (mCIMT) has been successfully used with children who have hemiplegia (weakness or paralysis on one side of the body.) mCIMT uses a removable cast during treatment and home exercise programs. It has been found that mCIMT can improve use, strength and coordination of a child's affected hand, and may also help improve speech and language skills. The goal of this project is to investigate whether combining mCIMT with speech therapy will enhance speech outcomes in children with cerebral palsy.

DETAILED DESCRIPTION:
Children with cerebral palsy (CP) often have hemiplegia, meaning only one side of the body is affected. They may have difficulty with daily tasks that require two hands. They may also have difficulty with speech and/or language. Constraint-induced movement therapy (CIMT) is a treatment that has been used to help improve children's performance of everyday activities and enhance their quality of life. CIMT uses a cast on the unaffected arm to encourage use of the affected hand. In traditional CIMT, a child wears a non-removable cast 24 hours a day for a duration of time. A more child-friendly version, modified constraint-induced movement therapy (mCIMT), uses a removable cast during treatment and home exercise programs. It has been found that mCIMT can improve use, strength and coordination of a child's affected hand. Preliminary studies have also shown some speech and language improvement in children with speech impairments who participated in mCIMT.

The goal of this project is to investigate whether combining mCIMT with speech and language treatment (SPT) will enhance speech outcomes when compared with SPT alone. We will examine (1) whether it is feasible and effective to deliver (SPT) and mCIMT simultaneously, and (2) whether providing mCIMT simultaneously with SPT leads to greater gains in speech-language outcomes than SPT alone? Such information could add valuable evidence-based treatment options for children with hemiplegia and comorbid speech-language deficits, change the way in which we plan patients' care, and help justify co-treating patients who get mCIMT. We hypothesize that forced use of the impaired limb in therapeutic tasks would have spread effects resulting in increased rate of speech-language improvement during treatment intervals when the patient is casted.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of Cerebral Palsy
* Hemiplegia
* Speech-Language Impairment
* English as primary language spoken in the patient's home
* Normal or corrected hearing and vision

Exclusion Criteria:

* Presence of co-morbid developmental disability (not including specific language impairment) which has an impact on cognition, sensory processing, and/or social-pragmatic function
* Non-corrected hearing loss as evidenced by audiology report, failure to pass a newborn hearing screening, and/or performance on pure-tone testing.
* Non-corrected vision impairments
* Weakness on both sides or neither side of the body
* Bilingual speakers or patients who speak languages other than English
* Previous history of CIMT or mCIMT within the past 6 months.

Ages: 15 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Probes | Up to 15 weeks
  Number of trained words and phrases produced during a treatment session.

SECONDARY OUTCOMES:
Mean Length of Utterance | Up to 15 weeks
  Average length of utterances produced during treatment sessions
Test of Early Language Development (TELD) | Up to 15 weeks
  Standardized assessment of spoken language skills
Goldman-Fristoe Test of Articulation-2 (GFTA-2) | Up to 15 weeks
  Standardized assessment of production of sounds in words

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Dayanidhi, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naylor CE, Bower E. Modified constraint-induced movement therapy for young children with hemiplegic cerebral palsy: a pilot study. Dev Med Child Neurol. 2005 Jun;47(6):365-9. doi: 10.1017/s0012162205000721. PMID 15934484
- [Background] Sigurdardottir S, Vik T. Speech, expressive language, and verbal cognition of preschool children with cerebral palsy in Iceland. Dev Med Child Neurol. 2011 Jan;53(1):74-80. doi: 10.1111/j.1469-8749.2010.03790.x. Epub 2010 Oct 11. PMID 21039439
- [Background] Allison KM, Reidy TG, Boyle M, Naber E, Carney J, Pidcock FS. Speech production gains following constraint-induced movement therapy in children with hemiparesis. J Pediatr Rehabil Med. 2017;10(1):3-9. doi: 10.3233/PRM-170405. PMID 28339405